CLINICAL TRIAL: NCT00825903
Title: The Effects of Exercise on Physiological and Psychological Parameters in an Asthmatic Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Kasee Hildenbrand, Assistant Professor, Washington State University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 10460
Record Dates: First submitted 2009-01-16; First posted 2009-01-21 (Estimated); Last update posted 2012-01-04 (Estimated); Status verified 2011-12

CONDITIONS: Asthma, Bronchial
Keywords: aquatic exercise; asthma
MeSH Terms: conditions — Asthma | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Aquatic based exercise
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Exercise 3 times each week for a total of 12 weeks. Each session is 50 min. in length.

SUMMARY:
Exercise has been shown to have extensive health benefits both in normally functioning adults as well as in adults with asthma. A program of regular aquatic exercise may have unique benefits in the asthmatic population because of the known aerobic capacity development typical of such programs, combined with the unique value of immersion-produced improvements in respiratory endurance and cardiac output. The purpose of this study is to explore the effects of a 12 week long aquatic endurance training program on several physiological and psychological parameters related to coronary heart disease and type II diabetes in an asthmatic population.

DETAILED DESCRIPTION:
The study will run from August 2008 to May 2009. Recruitment and screening of participants will occur from August to December 2008 for inclusion into the clinical trial. Prior to the clinical trial participants will have a one hour informational session to clearly present the study, obtain signed informed consent and set up fitness/blood appointments for data collection. Data collection will begin the first week of school in January. The 12-week exercise protocol will start the second week of school and continue through the middle of April. Research participants will not have any exercise session during spring break (March 16-20). Final data collection will occur during the last two weeks of school. Pre-treatment and post-treatment data collection will include a fitness assessment and blood draw. Medication usage for asthma will be monitored on a weekly basis thoughout the clinical trial. Physical activity will also be monitored monthly.

The screening session is a 30-minute session where research participants complete health/behavior questionnaires and a physiological measure of lung function. Information to be collected in the health/behavior questionnaires includes: demographic and behavioral/lifestyle variables (sex, race, age, smoking status, and medical history).

The fitness assessment will be 60 minutes in length. At the beginning of the session participants will complete a survey to assess state anxiety (State-Trait Anxiety Inventory - Trait version Form X-1; Spielberger, Gorsuch, & Lushene, 1970). Heart rate variability will be measured through the ventral placement of 3 electrodes placed on the subject's torso. The areas will be prepped by swabbing with alcohol and lightly scrubbing to remove dead skin. The electrodes will be held in place with a sticky disc and a strip of athletic tape. Heart rate and resting blood pressure will also be taken. Body composition will be assessed using the BodPod system. Research participants will sit in an enclosed capsule (bod pod) for three tests lasting approximately 40 seconds each. Lung function will be assessed using a spirometer to measure the maximal volume of air exhaled over a period of time after a maximal inhalation. To assess cardiorespiratory fitness research participants will complete a VO2 Max test. Participants will ride a bicycle ergometer for approximately 15-20 minutes moving through stages (including a 3 minute warm-up) with progressively higher resistance levels until maximum tolerance. After termination there is a cool-down/recovery period of approximately 3-4 minutes.

The blood draw session will take approximately 30 minutes and participants will be asked to fast (no food or drink) for 12 hours prior to blood draw. Upon check-in participants will complete a series of questionnaires assessing psychological variables stress (Perceived Stress Scale-14 item version Form X-1; Cohen, Kamarck & Mermelstein, 1983), depression (Center for Epidemiological Studies - Depression Scale; Radloff, 1977), and quality of life (Asthma Impact Survey; QualityMetric Health Outcomes Solutions, Lincoln, RI). The quality and quantity of sleep will also be assessed using the Pittsburgh Sleep Quality Index (Buysse, Reynolds, Monk, Berman, & Kupfer, 1989). Once questionnnaires are completed, participants will have their blood drawn by a certified phlebotomist. Three days after the blood draw particpants will be contacted by phone and questioned about current health status.

After the first week of pretreatment data collection, before the training sessions begin, research participants will undergo an explanation and training session to learn how to evaluate their own rate of perceived exertion (RPE). The water-based exercise programs are 3 times a week for 12 weeks. The exercise sessions will begin with a 10-minute warm up and end with a 5-minute cool down period. The conditioning portion of the exercise program will be shorter in duration with lower intensities at the beginning of the 12 weeks. There will be a progression to higher intensities for longer periods of time throughout the 12 weeks using recommendations from the American College of Sports Medicine. Exercise sessions will not exceed 50 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Medically diagnosed and medication managed asthmatics between the ages of 18-40

Exclusion Criteria:

* outside the age range of 18-40 years old, fear of water, diseases or conditions listed during screening process, or current smoker.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-09; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function | baseline and 12 weeks post

SECONDARY OUTCOMES:
Demographic information | baseline
Medical history | baseline
Smoking practices | baseline
Exercise practices | baseline and monthly
State Anxiety | baseline and 12 weeks post
Perceived Stress | baseline and 12 weeks post
Depression | baseline and 12 weeks post
Sleep - duration and quality | baseline and 12 weeks post
Quality of Life as related to asthma | baseline and 12 weeks post
Body composition | baseline and 12 weeks post
Cardiovascular fitness level- VO2 max | baseline and 12 weeks post
Resting Heart Rate | baseline and 12 weeks post
Heart Rate Variability and ECG | baseline and 12 weeks post
Serum cholesterol levels | baseline and 12 weeks post
Fasting blood glucose | baseline and 12 weeks post
Cortisol | baseline and 12 weeks post
Insulin | baseline and 12 weeks post
CRP | baseline and 12 weeks post
Homocysteine | baseline and 12 weeks post
Lipoprotein-Associated Phospholipase A2 (PLAC) | baseline and 12 weeks post
Medication usage | prior and throughout study
Exercise Adherence | throughout study
Resting blood pressure | baseline and 12 weeks post

CONTACTS AND LOCATIONS:
Overall Officials: Kasee J Hildenbrand, PhD, Principal Investigator — Washington State University
Locations (1):
- Washington State University, Pullman, Washington, United States